CLINICAL TRIAL: NCT00490529
Title: Phase 1-2 Study of a CpG-Activated Whole Cell Vaccine Followed by Autologous "Immunotransplant" for Mantle Cell Lymphoma
Brief Title: Phase 1-2 of a CpG-Activated Whole Cell Vaccine Followed by Autologous Immunotransplant for MCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ronald Levy (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Ronald Levy, Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-05089; LYMNHL0040-BMT212 (Other: OnCore); 96940 (Other: Stanford University Alternate IRB Approval Number); NCI-2011-00136 (Other: NCI Trial ID)
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma, Mantle-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ProMune; Transplantation; Rituximab; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CpG-MCL Vaccine (Experimental): An autologous anti-tumor vaccine.
  Interventions: Biological: CpG-MCL vaccine; Biological: PF-3512676; Procedure: Vaccine-primed T-cells; Procedure: Autologous hematopoietic stem cell transplant (HSCT); Drug: Rituximab; Drug: Standard induction chemotherapy; Drug: Cyclophosphamide; Drug: Filgrastim

INTERVENTIONS:
Biological: CpG-MCL vaccine — CpG-MCL vaccine is a vaccine prepared by co-culturing cells from the participant's mantle cell lymphoma suspension with 3 mcg/mL PF-3512676, then irradiated to 200 Gy. 1 x 10e8 CpG-MCL cells will be given as a subcutaneous injection.
  Other Names: CpG-activated, autologous tumor vaccine; Cytosine-Guanosine repeats (CpG)-mantle cell lymphoma (CpG-MCL vaccine)
Biological: PF-3512676 — PF-03152676 is a synthetic immunostimulatory, single-stranded oligodeoxynucleotide (oligo-DNA) moledule containing unmethylated cytosine and guanine (CpG) motifs. PF-03512676 acts as an agonist of human Toll-like receptor 9, leading to activation of antigen-presenting cells and a cascade of antitumor immune reactions.
  Other Names: CPG-7909
Procedure: Vaccine-primed T-cells — Vaccine primed T-cells are the post-vaccination leukapheresis harvest of peripheral blood mononuclear cells. Each collection is approx 1 x 10e10 CD3+ T-cells.
Procedure: Autologous hematopoietic stem cell transplant (HSCT) — Regular medical procedure
  Other Names: Autologous peripheral blood progenitor cell (PBPC) transplant; Autologous peripheral blood stem cell (PBSC) transplant
Drug: Rituximab — 375 mg/m² by infusion
  Other Names: Rituxan; hera
Drug: Standard induction chemotherapy — Patient-specific, regular medical care treatment as determined by treating oncologist
Drug: Cyclophosphamide — Regular medical care treatment to mobilize peripheral blood progenitor cell (PBPC)
  Other Names: Cytoxtan; Neosar; CYT; CTX; CPM
Drug: Filgrastim — Regular medical care treatment to mobilize peripheral blood progenitor cell (PBPC)
  Other Names: G-CSF; Neupogen

SUMMARY:
Mantle cell lymphoma (MCL) is a sub-type of non-Hodgkin's lymphoma (NHL) which is generally considered incurable with current therapy. Participants will receive an autologous vaccine against their individual lymphoma after undergoing stem cell transplantation. This vaccination may prolong the time which patients will stay in remission from their disease.

DETAILED DESCRIPTION:
Study treatment is a complex set of steps of research procedures and regular medical care. By using a participant's cancer cells as an immungen, the study hopes to improve freedom from molecular residual disease (MRD).

PRIMARY OBJECTIVE Freedom from molecular residual disease at 1-year post-autologous transplant.

SECONDARY OBJECTIVE Time To Clinical Progression (TTP)

This study has 2 research agents, PF-03152676 and CpG-MCL Vaccine.

PF-03152676 is a synthetic DNA molecule, 24 nucleotides in length with a nuclease-resistant phosphorothioate backbone. It is an immunostimulatory, single-stranded oligodeoxynucleotide (oligo-DNA) containing unmethylated cytosine and guanine (CpG) motifs and synthesized with a nuclease-resistant phosphorothioate backbone. PF-03512676 acts as an agonist of human Toll-like receptor 9, leading to activation of antigen-presenting cells and a cascade of anti-tumor immune reactions.

CpG-MCL Vaccine is the primary study agent. It is prepared by dissociating a participant's harvested tumor cells into a single-cell suspension, and culturing them with PF-03152676 for 72 hours at 37 degrees C, 5% CO2 to allow for up-regulation of antigen-presenting and co-stimulatory molecules, then irradiated to 200 Gy to destroy any remaining cancer propagating ability.

The study procedure is summarized as 12 steps, listed below.

* Step 1. Undergo excisional tumor biopsy or apheresis to obtain tumor cells, which will be used to generate the CpG-MCL vaccine .
* Step 2. Receive standard induction chemotherapy (regular medical care).
* Step 3. Once in remission, receive 3 vaccinations of CpG-MCL Vaccine over 3 weeks. With each CpG-MCL vaccination, a concurrent subcutaneous injection of PF-3512676 is administered as an adjuvant.
* Step 4. About 4 weeks later, receive rituximab 375 mg/m² to minimize any residual tumor.
* Step 5. Apheresis procedure to harvest the CpG-MCL Vaccine-primed T-cells. Each collection is ~1 x 10e10 CD3+ T-cells.
* Step 6. High-dose cytoxan and filgrastim to mobilize peripheral blood progenitor cell (PBPC).
* Step 7. Undergo separate apheresis procedure to harvest PBPC).
* Step 8. Receive myeloablative chemotherapy (regular medical care).
* Step 9. Receive PBPC infusion (also known as autologous hematopoietic cell transplant, AHCT).
* Step 10. Within 3 days of AHCT (but typically 1 day), receive infusion of CpG-MCL Vaccine-primed T-cells, followed within 1 hour by a with 4th vaccination with CpG-MCL Vaccine (1st booster vaccination).
* Step 11. After hematopoietic recovery, receive 5th vaccination with CpG-MCl (2nd booster vaccination).
* Step 12. Monitor participants for general health and disease status through at least 3 years.

ELIGIBILITY:
INCLUSION CRITERIA

* Newly-diagnosed with mantle cell lymphoma (MCL) with accessible disease site for excisional biopsy, OR have sufficient peripheral blood tumor to leukapherese ≥ 1.5 x 10e9 lymphoma cells in a single session
* Medically appropriate by standard clinical criteria to receive rituximab and standard induction chemotherapy and high-dose chemotherapy with autologous hematopoietic cell transplant (AHCT)
* HIV-negative
* Eastern Cooperative Oncology Group (ECOG) Performance Status, OR Karnofsky performance scale 50 to 100%
* Capable of providing informed consent

EXCLUSION CRITERIA

* Currently receiving immunosuppressive medications
* Severe psychological or medical illness
* Pregnant or lactating
* Unable to safely complete the study, at the discretion of the principal investigator

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-08; Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Levy, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brody JD, Goldstein MJ, Czerwinski DK, Levy R. Immunotransplantation preferentially expands T-effector cells over T-regulatory cells and cures large lymphoma tumors. Blood. 2009 Jan 1;113(1):85-94. doi: 10.1182/blood-2008-05-155457. Epub 2008 Sep 23. PMID 18812472
- [Result] Czerwinski DK, Brody J, Kohrt HE, et al. "Immunotransplant Expands Vaccine Induced Memory T cell Responses In Patients With Mantle Cell Lymphoma." Blood. 2013;122(21)1816.
- [Result] Chu MP, Brody J, Kohrt HE, et al. "Phase I/II Clinical Trial of CpG Activated Whole Cell Vaccine in Mantle Cell Lymphoma (MCL): Results in Safety and Efficacy from Planned Interim Analysis Blood." Blood. 2015;126(23)
- [Result] Frank MJ, Khodadoust M, Chu M, et al. "Phase I/II Clinical trial of an activated whole tumor cell vaccine followed by transfer of immune T cells in patients with Mantle Cell Lymphoma." Hematological Oncology). 7 June 2017, https://doi.org/10.1002/hon.2438_72.
- [Derived] Frank MJ, Khodadoust MS, Czerwinski DK, Haabeth OAW, Chu MP, Miklos DB, Advani RH, Alizadeh AA, Gupta NK, Maeda LS, Reddy SA, Laport GG, Meyer EH, Negrin RS, Rezvani AR, Weng WK, Sheehan K, Faham M, Okada A, Moore AH, Phillips DL, Wapnir IL, Brody JD, Levy R. Autologous tumor cell vaccine induces antitumor T cell immune responses in patients with mantle cell lymphoma: A phase I/II trial. J Exp Med. 2020 Sep 7;217(9):e20191712. doi: 10.1084/jem.20191712. PMID 32558897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Some participants started study procedures, but did not receive the intended study treatment.
Period: Completed Pre-CpG-MCL Vaccine Procedures
Arm/Group | CpG-MCL Vaccine
Started | 59
Completed | 48
Not Completed | 11
Not completed — Death | 4
Not completed — Withdrawal by Subject | 4
Not completed — Withdrawn, AHCT not suitable treatment | 1
Not completed — Withdrawn, chemo not suitable treatment | 1
Not completed — Withdrawal due to insurance refusal | 1
Period: Treatment With CpG-MCL Vaccine
Arm/Group | CpG-MCL Vaccine
Started | 48
Completed | 47
Not Completed | 1
Not completed — Received vaccine, did not receive AHCT | 1

BASELINE CHARACTERISTICS:
Population: Includes all participants that started study procedures. Prospective participants that consented but did not receive any research procedures are not included.
Arm/Group | CpG-MCL Vaccine
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 54
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Molecular Residual Disease (MRD) Post-autologous Stem Cell Transplant (ASCT)
Description: Molecular residual disease (MRD) is defined as detection in blood samples by the ClonoSEQ test of the (11;14) (q13;q32) gene translocation. It is considered positive if a tumor-specific VDJ sequence is detected in the peripheral blood cells by Ig-HTS at a frequency of greater or equal to 1 molecule per 10,000 input leukocyte equivalents of DNA within 1 year post-autologous stem cell transplant (ASCT). The outcome will be reported as number and percent of participants that maintain MRD-negative status (ie, 1-year freedom from MRD). This outcome is reported as a number without dispersion.
Time Frame: 12 months
Population: Only participants for which molecular residual disease (MRD) disease status assessments were available are included.
Measure: Count of Participants; unit: Participants
Groups:
- CpG-MCL Vaccine: An autologous anti-tumor vaccine.
  CpG-MCL vaccine: CpG-MCL vaccine is a vaccine prepared by co-culturing cells from the participant's mantle cell lymphoma suspension with 3 mcg/mL PF-3512676, then irradiated to 200 Gy. 1 x 10e8 CpG-MCL cells will be given as a subcutaneous injection.
  PF-3512676: PF-03152676 is a synthetic immunostimulatory, single-stranded oligodeoxynucleotide (oligo-DNA) moledule containing unmethylated cytosine and guanine (CpG) motifs.
  Vaccine-primed T-cells: Vaccine primed T-cells are the post-vaccination leukapheresis harvest of peripheral blood mononuclear cells. Each collection is approx 1 x 10e10 CD3+ T-cells.
  Autologous hematopoietic stem cell transplant (HSCT): Regular medical procedure
  Rituximab: 375 mg/m² by infusion
  Standard induction chemotherapy: Patient-specific, regular medical care treatment as determined by treating oncologist
  Cyclophosphamide: Regular medical care treatment to mobilize peripheral blood progenitor cell (PBPC)
Arm/Group | CpG-MCL Vaccine
Number analyzed (Participants) | 45
Participants | 41

2. Secondary Outcome: Time-to-progression (TTP)
Description: Time-to-progression (TTP) is measured from the time of autologous stem cell transplantation (ASCT) until the cancer progresses or relapses. Progression is assessed based on CT imaging per the Cheson Criteria (2008). Progression per the Cheson Criteria is defined as having occurred when the sum of tumor lesion dimensions is ≥ 150% of the baseline value. The outcome is reported as the median with 95% confidence interval, as determined by Kaplan-Meier analysis and log-rank test.
Time Frame: 7.7 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | CpG-MCL Vaccine
Number analyzed (Participants) | 47
years | 6.9 [5.92 to NA] — The upper end of the 95% confidence interval was not reached.

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) rate is reported as number and percentage of participants remaining alive the date of transplant through each year, up to 5 years (reported as a number without dispersion).
Time Frame: After 1, 2, 3, 4, and 5 years
Population: Only participants that received the CpG-MCL Vaccine are included.
Measure: Count of Participants; unit: Participants
Arm/Group | CpG-MCL Vaccine
Number analyzed (Participants) | 48
Participants
  OS after 1 year | 42
  OS after 2 year | 33
  OS after 3 year | 27
  OS after 4 year | 19
  OS after 5 year | 13

4. Secondary Outcome: Detection of Tumor-specific CD8-positve Memory T-cells Before and After Vaccination
Description: Anti-tumor T-cell immune responses were evaluated by an in vitro evocative test on their peripheral blood mononuclear cell (PBMCs) before and after vaccination, as assessed by measurement of intracellular cytokines and/or intracellular perforin/granzyme in CD8+ T-cells, and/or CD137 induction on CD4+ T-cells. PBMCs were co-cultured with CpG-activated autologous MCL tumor cells and evaluated for tumor-specific immune responses as measured by CD137 expression on their T cells. The outcome is reported as the number of participants for whom tumor-specific memory CD8 cells were detected at baseline and after vaccination and transplant (numbers without dispersion).
Time Frame: Baseline and after vaccination and transplant, approximately 5 years
Population: Only participants for which both baseline and post-transplant assessments were available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | CpG-MCL Vaccine
Number analyzed (Participants) | 35
Participants
  At Baseline | 31
  After Transplant | 14

5. Secondary Outcome: Detection of Tumor-specific CD4-positve T-cells Before and After Vaccination
Description: Anti-tumor T-cell immune responses were evaluated by an in vitro evocative test on their peripheral blood mononuclear cell (PBMCs) before and after vaccination, as assessed by measurement of intracellular cytokines and/or intracellular perforin/granzyme in CD8+ T-cells, and/or CD137 induction on CD4+ T-cells. PBMCs were co-cultured with CpG-activated autologous MCL tumor cells and evaluated for tumor-specific immune responses as measured by CD137 expression on their T cells. The outcome is reported as the number of participants for whom tumor-specific memory CD4 cells were detected at baseline and after transplant (numbers without dispersion).
Time Frame: Baseline and after vaccination and transplant, approximately 5 years
Population: Only participants for which both baseline and post-transplant assessments were available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | CpG-MCL Vaccine
Number analyzed (Participants) | 35
Participants
  At Baseline | 20
  After Transplant | 14

ADVERSE EVENTS:
Time Frame: 3 months
Description: The study has 2 stages, ie, procedures preceding vaccine administration + the vaccine treatment period.
  * All cause mortality includes the entire subject population (ie, both pre-vaccine period and actual treatment period).
  * Serious Adverse Events and Other (Not Including Serious) Adverse Events information includes only the participants that received the vaccine and transplant (actual study treatment period).
Arm/Group | CpG-MCL Vaccine
All-Cause Mortality (participants affected / at risk) | 19/59
Serious Adverse Events (participants affected / at risk) | 31/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CpG-MCL Vaccine (N=48)
Hemorrhage, CNS, Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, Graft failure (Blood and lymphatic system disorders) | 1 (1)
Infection, dental abscess (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Investigations) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Supraventricular and nodal arrhythmia (Vascular disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2)
Death Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12)
Burn (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CpG-MCL Vaccine (N=48)
Pain Joint (Arthalgia) (Musculoskeletal and connective tissue disorders) | 16 (35)
Phantom sensations (sensitivity/crawly feeling on skin) (Psychiatric disorders) | 2 (2)
Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 4 (7)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Distension/bloating Abdominal (Gas/indigestion) (Gastrointestinal disorders) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3)
Fatigue (General disorders) | 25 (53)
Fever (General disorders) | 29 (63)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Flu-like syndrome: General (General disorders) | 4 (4)
Head/Headache (Nervous system disorders) | 16 (26)
Heartburn/dyspepsia (Gastrointestinal disorders) | 5 (6)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Imsomnia (Nervous system disorders) | 2 (3)
Induration (Skin and subcutaneous tissue disorders) | 14 (21)
Metapneumovirus (Infections and infestations) | 1 (1)
Injection site reaction/extravasation changes: Erythema (General disorders) | 47 (123)
Injection site reaction/extravasation changes: Pain (General disorders) | 19 (39)
Injection site reaction/extravasation changes: Swelling (General disorders) | 24 (63)
Injection site reaction/extravasation changes: Warmth (General disorders) | 17 (35)
Joint Function (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytes count low (Blood and lymphatic system disorders) | 3 (3)
Lymphocytes count low (Blood and lymphatic system disorders) | 1 (1)
Mucositis/Stomatitis (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (62)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Neutrophils/granulocytes count low (Investigations) | 4 (4)
Other: Granuloma (Skin and subcutaneous tissue disorders) | 1 (1)
Other: thinning/fragile skin (Skin and subcutaneous tissue disorders) | 2 (2)
Platelets count low (Blood and lymphatic system disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritis/Itching (Skin and subcutaneous tissue disorders) | 12 (15)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 6 (6)
Rigors/Chills (General disorders) | 22 (45)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Voice changes/dysarthia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight Loss (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT00490529/Prot_SAP_000.pdf